CLINICAL TRIAL: NCT06304129
Title: Threshold Values and Diagnostic Performance of Plasma Biomarkers of Alzheimer's Disease Compared With CSF Markers
Brief Title: Diagnostic Performance of Plasma Biomarkers of Alzheimer's Disease Compared With CSF Markers
Acronym: PLASM-ALZ
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Thérèse Jonveaux (Unknown); Laure Joly (Unknown); Lucie Hopes (Unknown); Maia Simon (Unknown); Franck Schreiner (Unknown)
Responsible Party: Principal Investigator, Catherine MALAPLATE, Dr, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-A00709-36
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-09

CONDITIONS: Alzheimer Blood Biomarkers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood ponction (Experimental): All patients are in the experimental group
  Interventions: Diagnostic Test: Blood ponction

INTERVENTIONS:
Diagnostic Test: Blood ponction — Blood ponction

SUMMARY:
.The goal of this interventional study is to estimate the diagnostic performance of plasma biomarkers of interest (Aβ40 and Aβ42, P-Tau and NFL), enabling discrimination between patients with and without a pathophysiological AD process. The main questions it aims to answer are:

* to define a threshold value for each of the plasma,
* to describe the correlations between the plasma biomarkers of interest and the other biological analyses performed as part of care, in particular triglyceridemia, cholesterolemia, glycemia and proteinemia,
* to describe biomarker results in relation to comorbidities, in particular dyslipidemia and diabetes
* to describe the final diagnosis and results obtained for plasma biomarkers, for patients with intermediate results according to the A/T/N classification (A-/T+ or A+/T-) Participants will be selected among patients undergoing lumbar puncture for the differential diagnosis of AD at Nancy University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 18 or over
* Person affiliated to a social security scheme or beneficiary of such a scheme
* Person who has received full information on the organization of the research and has signed an informed consent form
* Person whose care requires a lumbar puncture to measure markers of Alzheimer's disease

Exclusion Criteria:

* Adult subject to a legal protection measure (guardianship, curatorship, safeguard of justice)
* An adult unable to give consent
* Persons deprived of their liberty by judicial or administrative decision
* Persons under psychiatric care under articles L. 3212-1 and L. 3213-1.
* Pregnant, parturient or breast-feeding women
* Persons staying in a health or social establishment for purposes other than research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Estimated)
Dates: Start 2024-04-02 (Estimated); Primary Completion 2026-01-02 (Estimated); Study Completion 2026-09-02 (Estimated)

PRIMARY OUTCOMES:
Aβ40 and Aβ42, P-Tau, Tau and NFL | 2 years
  Peptides Aβ40 and Aβ42, P-Tau and NFL, assayed in plasma. Peptides Aβ40 and Aβ42, Tau and P-Tau assayed in CSF

SECONDARY OUTCOMES:
Sensitivity/specificity | 2 years
  sensitivity, specificity, positive predictive value and negative predictive value of the plasma biomarkers of interest (Aβ40 and Aβ42, P-Tau and NFL) according to the defined threshold value, with reference to the A/T/N classification
Co-mobidity | 2 years
  results of assays for plasma biomarkers of interest (Aβ40 and Aβ42, P-Tau and NFL) in subgroups of patients with co-morbidities (notably dyslipidemia, diabetes)
Final diagnosis | 2 years
  final diagnosis selected according to criteria used in clinical practice (based on a multidisciplinary approach including analysis of biological results) and measurement of plasma biomarkers (Aβ40 and Aβ42, P-Tau and NFL) in the subgroup of patients with intermediate results according to the A/T/N classification (A-/T+ or A+/T-)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Malaplate, PhD, PharmD, Principal Investigator — CHRU Nancy
Locations (1):
- CHRU De Nancy, Nancy, Grand Est, France

IPD SHARING:
Plan to Share IPD: Undecided